CLINICAL TRIAL: NCT04980729
Title: A Novel Positioning Navigation Template for Accurately and Precisely Assisting the Placement of Modular Hemipelvic Endoprostheses for Patients Undergoing Pelvic Bone Tumor Resection: A Retrospective Cohort Study
Brief Title: A Positioning Navigation Template for Assisting the Placement of Modular Hemipelvic Endoprostheses for Patients Undergoing Pelvic Bone Tumor Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-453
Record Dates: First submitted 2021-05-30; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-05

CONDITIONS: Pelvic Tumor
Keywords: Pelvic tumor; Acetabular reconstruction; Navigation template; Hip rotation center; Placement in situ
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a "Retrospective Cohort Study" through retrospectively collecting patients undergoing acetabulum reconstruction after pelvic tumor resection. The patients were interfered with or without the acetabular navigation template during the hip reconstruction process.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the template-guided group (Experimental): In the template-guided group (n = 10), a navigation template was designed and applied to assist acetabular reconstruction using a modular hemipelvic prosthesis.
  Interventions: Device: Acetabular reconstruction after tumor resection.
- the traditional operation group (Active Comparator): In the traditional operation group (n = 14), acetabulum was manually reconstructed using a modular hemipelvic prosthesis by the surgeon's experience.
  Interventions: Device: Acetabular reconstruction after tumor resection.
- the validation group (Sham Comparator): In the validation group (n = 12), patients undergoing periacetabular puncture or curettage without acetabulum reconstruction.
  Interventions: Device: Acetabular reconstruction after tumor resection.

INTERVENTIONS:
Device: Acetabular reconstruction after tumor resection. — In the template-guided group (n = 10), a navigation template was designed and applied to assist acetabular reconstruction. In the traditional operation group (n = 14), the patients underwent the same surgery but without the navigation template. To compare the displacement of the hip rotation center before and after surgery between the two groups, an innovative method based on pelvic CT was developed and a validation group of cases was used to assess the effectiveness of this measurement approach. In the validation group (n = 12), patients undergoing periacetabular puncture or curettage without hip joint reconstruction were included. The displacements for the validation group were calculated and compared with 0 cm, the theoretical value. Subsequently, the displacements between the template-guided group and the traditional operation group were compared.

SUMMARY:
Background:

Acetabular reconstruction in situ after extensive pelvic resection is technically challenging because the significant loss of bone stock and bony landmarks. The aim of the present study was to investigate the feasibility of an individualized navigation template for acetabular reconstruction following pelvic malignancy resection.

Methods:

This retrospective cohort study included patients who underwent type II or II+III pelvic tumor resection and reconstruction using a modular hemipelvic prosthesis. In the template-guided group (n = 10), a navigation template was designed and applied to assist acetabular reconstruction. In the traditional operation group (n = 14), the patients underwent the same surgery but without the navigation template. To compare the displacement of the hip rotation center before and after surgery between the two groups, an innovative method based on pelvic CT was developed and a validation group of cases was used to assess the effectiveness of this measurement approach. In the validation group (n = 12), patients undergoing periacetabular puncture or curettage without hip joint reconstruction were included. The displacements for the validation group were calculated and compared with 0 cm, the theoretical value. Subsequently, the displacements between the template-guided group and the traditional operation group were compared.

ELIGIBILITY:
Inclusion Criteria:

1. All the patients diagnosed with a pelvic tumor；
2. Underwent limb salvage surgery following type II or II+III pelvic resection；
3. Acetabulum reconstruction using a modular, titanium hemipelvic prosthesis.

Exclusion Criteria:

1. A lack of postoperative CT images;
2. Having undergone revision surgery or noninitial/primary resection;
3. unable to calculate the hip displacement by the specific measurement method we proposed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Compare the change of acetabular rotation center before and after surgery between the template-guided group and the traditional operation group. | "through study completion, an average of 2 years"
  Compare the change of acetabular rotation center (the displacement displayed in centimeters) before and after surgery between the template-guided group and the traditional operation group based on preoperative and postoperative CT images.

CONTACTS AND LOCATIONS:
Overall Officials: Nong Lin, Study Director — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Donghua Huang, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No